CLINICAL TRIAL: NCT05316194
Title: Minimal Clinically Important Changes in Digitally Delivered Osteoarthritis Treatment
Brief Title: Minimal Clinically Important Changes in Osteoarthritis Treatment
Status: Completed | Type: Observational
Sponsor: Joint Academy (Industry)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: MIC in OA
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: Osteoarthritis; Minimal Clinically Important Change; Responder; Exercise; Telehealth; Digital; Knee; Hip; Treatment failure; Patient acceptable symptom state
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Osteoarthritis; Motor Activity | interventions — Papaverine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participation in digital OA treatment: All participants that have participated in a digitally delivered first-line treatment program (Joint Academy) for hip or knee OA until May 2022.
  Interventions: Other: Digital treatment for hip and knee osteoarthritis

INTERVENTIONS:
Other: Digital treatment for hip and knee osteoarthritis — The program is an app-based version of the Swedish face-to-face management program for OA "Better management of patients with OsteoArthrits" and includes weekly educational sessions, individualized exercises and a possibility to chat asynchronously with a physical therapist during the entire duration of the program.

SUMMARY:
To assess minimal clinically important change, cut-offs for treatment failure and patient acceptable symptom state for pain and patient-reported function and quality of life in persons with hip or knee osteoarthritis, participating in digitally delivered first-line education and exercise treatment.

DETAILED DESCRIPTION:
Patient-reported outcome measures (PROMs) are consistently recommended as the primary end-point in clinical trials evaluating treatment effects in different medical conditions. For a meaningful interpretation of the PROMs used, three different approaches have been proposed; The Minimal Important Change (MIC), which is the smallest change in scores that represents an important improvement for the patient, i.e., the patient is feeling better, the Patient Acceptable Symptom State (PASS), which represents patients that consider their current status as acceptable, i.e., the patient is feeling good and Treatment Failure (TF), which represents patients that consider their state so unsatisfactory that they think the treatment has failed, all based on relevant anchor questions. Previous research in patients with anterior cruciate ligament (ACL) injury and femoroacetabular impingement reveals that feeling better is not necessarily the same as feeling good and reporting only the MIC (or mean change) may overestimate the results, stressing the need for including different measures of improvement to evaluate treatment effects on PROMs. The MIC, PASS and TF for persons undergoing digital treatment for hip or knee osteoarthritis are not yet determined. In this retrospective register-based study we will define MIC, PASS and TF in pain and patient-reported function and quality of life, using anchor-based questions, for persons participating in digital first-line treatment for hip and knee OA. In addition, we will use these thresholds to establish the proportion of patients reaching MIC and/or PASS or reporting TF, separate for persons with hip and knee OA.

Statistical analysis:

For MIC calculations, participants will be categorized as "importantly improved" if they answered "Better an important improvement" or "Somewhat better but enough to be an important improvement" to the anchor questions for KOOS/HOOS and NRS. MIC for an important improvement will then be calculated using the predictive modeling method (MICpred), adjusting for the proportion of improved patients.

The MICpred method will also be used to calculate the post score (i.e., 3, 6, 9 and 12 months) for KOOS/HOOS-scores and NRS-scores for participants that have responded "Yes" to the PASS or TF anchor question, respectively. The proportion of participants reaching the cut-offs of MIC, PASS and TF for the KOOS/HOOS and NRS, will then be calculated separately for participants with knee and hip OA.

Subgroup analyses on the effect of sex, age and baseline symptoms (depending on data distribution to ensure we will have an adequated sample size also in subgroups) on MIC, PASS and TF will also be performed using the MICpred method

ELIGIBILITY:
Data for all participants enrolled in the program until May 2022, and have given their written informed consent, will be extracted from the digital treatment register.

Inclusion criteria will be; i) diagnosed hip or knee OA ii) provided answer for KOOS/HOOS questionnaires and/or NRS pain at baseline and any of the follow-ups, i.e., 3, 6, 9 and/or 12 months.

Exclusion criteria: none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants join the digital OA treatment program via online advertisements and campaigns placed on search engines and social networks, or by recommendations by their local care provider. Radiographic and or clinical diagnosis of hip or knee OA from a physical therapist or physician (95% of all patients in previously published studies). Individuals without a prior diagnosis had clinical OA confirmed by an orthopaedic surgeon or physiotherapist via telephone (diagnosis according to NICE criteria and Swedish National Guidelines, and confirming the absence of any red flag symptoms), or if deemed necessary were recommended to seek face-to-face care before inclusion in the programme.
  From October 1st 2021, all patients should have undergone a physical examination by doctor or physiotherapists before being able to enter the treatment.
Sampling Method: Non-Probability Sample
Enrollment: 11708 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Joint pain | 3 - 12 months
  Joint pain will be measured with the NRS-scale. NRS comprises an 11-point scale where 0 indicates no pain and 10 indicates the worst possible pain during the last week
KOOS/HOOS-12 | 3-12 months
  The Knee injury and Osteoarthritis Outcome Score (KOOS-12)(knee OA) and the Hip injury and Outcome Score (HOOS)(hip OA) will be used for evaluating knee/hip function and quality of life. The KOOS/HOOS-12 are short versions of the original KOOS/HOOS questionnaires and includes 12 items measuring knee/hip pain, physical function and knee/hip-related quality of life. All items are scored from 0-4. The scores will then be normalized to a score from 0-100 for each domain (pain, function and quality of life) as well as a total score of all three domains where 0 indicates extreme problems and 100 indicates no problems.
MIC | 3 - 12 months
  The MIC associated with KOOS/HOOS-12/NRS scores will be calculated using domain specific anchor questions; NRS and KOOS/HOOS pain: How is your joint pain now compared with prior to your participation in the treatment? KOOS/HOOS function: How is your ability to perform daily activities now, compared with prior to your participation in the treatment? (sitting, standing, walking, stairs, putting on/taking off socks, household work)? KOOS/HOOS QoL: How is your quality of life in relation to your knee now, compared with prior to your participation in the treatment? (trust in knee, lifestyle, how often you think of your knee)? With the following response option; Better, an important improvement/ Somewhat better but enough to be an important improvement/ Very small change, not enough to be an important improvement/About the same/Very small change, not enough to be an important deterioration/Somewhat worse, but enough to be an important deterioration/Worse, an important deterioration
Patient acceptable symtom state (PASS) | 3 - 12 months
  The following question will be asked (yes/no); Considering your knee/hip function, do you feel that your current state is satisfactory? You should take all activities during your daily life, sport and recreational activities, your level of pain and other symptoms, and also your knee/hip- related quality of life into account.
Treatment failed (TF) | 3 - 12 months
  The following question will be asked (yes/no): If you answered "No" to the previous question, would you consider your current function as being so unsatisfactory that you think the treatment has failed?

CONTACTS AND LOCATIONS:
Overall Officials: Leif E Dahlberg, Study Director — Arthro Therapeutics
Locations (1):
- Arthro Therapeutics, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No
IPD will only be shared between the researchers working with this project. According to the European General Data Protection Regulation (GDPR) we cannot legally share IPD outside of this project.